CLINICAL TRIAL: NCT06832033
Title: Effects of a Concurrent Physical Exercise Program in Patients Undergoing Atrial Fibrillation Ablation on Fibrillation Burden, Cardiac Morphology and Function, Physical Fitness, Physical Activity, Body Composition and Quality of Life.
Brief Title: Concurrent Training in Patients Undergoing Atrial Fibrillation Ablation.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marcos Echevarría (Other)
Responsible Party: Sponsor-Investigator, Marcos Echevarría, Sponsor-Investigator, Universidad de Zaragoza
Organization: Universidad de Zaragoza (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PI24/174
Record Dates: First submitted 2025-01-29; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-01

CONDITIONS: Atrial Fibrillation (AF); Physical Exercise; Physical Activity; Physical Fitness; Sleep; Quality of Life; Electrocardiogram; Echocardiogram
MeSH Terms: conditions — Atrial Fibrillation; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention)
- Training group (Active Comparator): This group carried out a concurrent physical exercise intervention for 12 weeks
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — 12 weeks of concurrent training, which is understood as a combination of strength and aerobic exercises, not necessarily in the same training session. The weekly frequency will be 3 times per week. The aerobic component of the session will last between 30 and 50 minutes (increasing as the weeks go by) and the strength work will be made up of 8 exercises (3 upper body and 5 lower body). The intensity of the training will be individualized and always moderate.
  Other Names: Concurrent training; Physical exercise
  Arms: Training group

SUMMARY:
Atrial fibrillation (AF) is an irregular and often very fast heart rhythm, is considered the most common sustained cardiac arrhythmia in adults worldwide, and its incidence and prevalence are increasing. Currently, the estimated prevalence of AF in adults is 2-4%, and is projected to increase 2.3-fold.

AF is associated with increased morbimortality and other comorbidities (hypertension diabetes etc.) which places a significant burden on the patient himself, social health and also on health and social care expenditure.

The European Society of Cardiology proposes an integrated ABC model (A: Anticoagulation, B: main symptom management, C: optimization of comorbidities and cardiovascular) and within this model, catheter ablation (B) is considered one of the main treatments to control AF symptoms; physical activity (C) is considered one of the modifiable health risk factors and is considered within a lifestyle intervention together with weight loss.

Catheter ablation of AF is currently the treatment of choice for paroxysmal AF. It uses small burns or frostbite to cause some scarring inside the heart to help interrupt the electrical signals that cause the irregular heartbeat. It is a safe procedure that has been shown to be more effective than treatment with antiarrhythmic drugs in reducing the arrhythmic burden and, therefore, the morbidity and mortality associated with the pathology.

Many studies have demonstrated the beneficial effects of moderate physical activity and physical exercise on cardiovascular health. However, there is still controversy as to whether physical activity is associated with an increased risk of AF in the general population; while some studies report a decreased risk of AF, others suggest an increase or that there is no evidence of an association between AF and physical activity.

Few studies have yet focused on the effects of physical activity in those subjects who have undergone catheter ablation. Studies that have evaluated physical activity with questionnaires associate it, when of moderate or high intensity, with lower recurrence of AF and lower incidence of serious events. It is true that the practice of regular and controlled physical exercise is a recognized part of the comprehensive care of patients with coronary heart disease (patients whose heart has difficulty receiving blood), and exercise is systematically identified as a central element of their rehabilitation. However, to date there is no similar approach for AF ablation patients.

Given the current situation of the subject of interest, the main objective of this project is to study the influence of a physical exercise program in patients undergoing catheter ablation of AF on different morphological and physiological variables of the heart, levels of physical activity and quality of life of patients. Investigators intend to recruit 120 participants, who will be randomly and equally distributed into a group that will perform a physical exercise intervention and a control group that will not perform any type of intervention. Participation in the study will not disrupt the normal practice of the health care system with these patients.

DETAILED DESCRIPTION:
This is a randomized, controlled trial. The study will be conducted in collaboration with researchers from the GENUD (Growth Exercise NUtrition and Development) and BSICoS (Biomedical Signal Interpretation and Computational Simulation) research groups at the University of Zaragoza (Spain), and also with the Hospital Clínico Universitario Lozano Blesa, Zaragoza (Spain), specifically with the arrhythmia department of the cardiology service of that hospital.

The main objective of the study is to study the effect of physical exercise in people who have undergone atrial ablation at least one year ago on AF recurrence, heart morphology and function, level of physical activity, sleep quality, physical condition, quality of life, and hospitalization or adverse events. In addition, investigators also aim to assess gender differences in response to physical exercise after atrial ablation on the above-mentioned variables. Due to the characteristics of the project, insurance has been contracted to cover possible risks that may be contemplated during training and evaluations.

The first phase of the study corresponds to the recruitment of subjects and will be carried out among patients in the Arrhythmia Unit of the Hospital. All patients who have been undergoing catheter ablation as a medical treatment for AF for one year will be invited to participate and all those who wish to participate in the study must complete the informed consent form. Therefore, the incorporation of participants in the study will be periodic (weekly and/or monthly) and "drop-by-drop".

The subjects who will participate in the study will be patients, women and men, over 18 years of age, who underwent catheter ablation as medical treatment for AF and who currently have no recurrence of this arrhythmia. The inclusion and exclusion criteria are detailed in the corresponding section.

To calculate the sample size, a statistical power analysis was performed through the G*Power program with the following input parameters to obtain the effect of time: effect size (f = 0.25), type I error (α = 0.05), power level or type II error (0.95), number of measurements (3: pre-, post-ablation and follow-up). Our analysis revealed a total sample size of 54 individuals per group. Based on the previous years' care activity, the investigators expect to recruit at least 60 patients for each group (intervention and control) to guarantee the number of 54, considering a dropout around 10%.

All participants (both groups) will be evaluated at 3 points in time. The first evaluation will be at the time of recruitment, prior to the start of the physical exercise intervention (month 0), to determine the patient's initial condition. The second evaluation will take place after the end of the intervention (month 3), to study the effects of physical exercise and the last one 6 months after recruitment, to assess the detraining of the intervention group and continue with the follow-up of the control group.

All assessments will consist of two days of measurements. One day will include physical fitness, physical activity, body composition and quality of life questionnaires and the other day will include cardiac assessment by echocardiogram and electrocardiogram. Each of the measurements is mentioned below (the measures are described in the corresponding section):

* Body composition.
* Electrocardiogram (ECG).
* Echocardiogram.
* Objective physical activity.
* Sleep analysis.
* Muscle strength.
* Cardiorespiratory capacity.
* Quality of life.
* Assessment of atrial fibrillation load.

The experimental design of the project is a randomized controlled trial where subjects will be assigned to one of two groups randomly defined using the randomizer.org website, considering sex and age: (a) control group, which will receive usual medical care and (b) experimental group, which will carry out a training program described below.

The intervention group will carry out a concurrent training program for 12 weeks, designed based on the scientific evidence currently available and following the latest recommendations (year 2023) for the diagnosis and management of AF from the American College of Cardiology (ACC) and the American Heart Association (AHA). During the 12 weeks of training (3 months) the weekly frequency will be 3 days per week. The duration of the sessions will increase progressively from week 1 to week 4. The sessions consist of resistance and aerobic training, and are divided into warm-up, resistance training with free weights (8 exercises, 3 for the lower body and 5 for the upper body), aerobic training on a cycle ergometer and a cool-down with stretching. Aerobic training will increase in duration from week 1 (30 min/day) to week 5 (50 min/day), following the principle of training progression. The same will be done with resistance work, being carried out once a week during the first 4 weeks and twice a week from weeks 5 to 12, adjusting the workloads individually based on the patient's progression.

The intensity of the training will be moderate and always individualized, based on the theoretical maximum heart rate (HRmax) calculated with the equation of Gellish et al. [207-(0.7*age)] for aerobic work (64-74% FCmax) and in repetitions in reserve (RIR) for resistance work (4-6). Overall, the perceived sense of effort is intended to be around 3-4 on the modified Borg scale (0-10). To perform a subsequent analysis of adherence to the physical exercise program by these patients, an individual attendance record will be made at the training sessions.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years
* Undergoing catheter ablation as medical treatment for AF at least one year prior to enrollment.

Exclusion Criteria:

* Patients who do not sign the informed consent for participation in the study.
* Severe atrial dilatation.
* Structural heart disease.
* Pathology that prevents the normal practice of intervention with physical exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Atrial fibrillation burden | 6 months
  By subcutaneously implanting an insertable Holter device, the exact time in AF can be accurately quantified, since this type of device continuously monitors the heart rhythm throughout its battery life (3 years). This allows all subclinical and clinical AF episodes and their duration to be recorded.
Echocardiogram | 6 months
  It will be performed by a single observer with a Vivid iQ model echocardiograph following the latest recommendations.
Cardiorespiratory capacity | 6 months
  A 6-minute walking test will be performed to assess the subjects' cardiorespiratory capacity.

SECONDARY OUTCOMES:
Body composition | 6 months
  Bioimpedance. A bioimpedance analyzer (TANITA MC-780) will be used to estimate fat mass.
Body composition | 6 months
  Bioimpedance. A bioimpedance analyzer (TANITA MC-780) will be used to estimate fat-free mass (muscle and bone mass).
Electrocardiogram (ECG) | 6 months
  Description and study of the ECG P wave, obtained from both single leads and combined information from multiple leads.
Electrocardiogram (ECG) | 6 months
  Study of heart rate variability (HRV) from the index of standard deviation of NN intervals (SDNNN).
Electrocardiogram (ECG) | 6 months
  Study of heart rate variability (HRV) from the root mean square of successive differences (RMSSD).
Objective physical activity | 6 months
  An Axivity X6 triaxial accelerometer (Newcastle upon Tyne, UK) will be used, which will be worn by the subject on the non-dominant hand for two weeks 24h a day. The recording frequency will be at 100Hz. The files will be analyzed through R-4.3.2 version of R software (http://cran.r-project. org), making use of the GGIR 3.0.5 package. The following variables will be generated and computed for all valid days: average acceleration (mg); total time in physical activity of moderate or vigorous intensity classified according to the cut-off point of 100 mg; the intensity gradient; the acceleration or intensity above which the X most active minutes are accumulated in the day (Mx, mg): M480, M120, M60, M30, M15, M10, M5, M2.
Sleep analysis | 6 months
  The R work package GGIR also allows for extracting sleep analysis information from data collected with accelerometers. Time periods with low variability in the accelerometer z-angle (i.e. <5° in 5 minutes) will be used and are defined as periods of sustained inactivity. Periods of sustained inactivity within these hours will be classified as sleep time. Data will be obtained on: sleep onset and end times, periods of wakefulness after sleep onset, and sleep efficiency.
Muscle strength | 6 months
  A hand-held dynamometer (TAKEY TKK-5401) will be used to measure handgrip strength. Two maximum strength measurements will be taken for each limb, in a bipedal position and with the arm extended and separated from the body. To evaluate lower body strength, the sit-to-stand test of 5 repetitions will be performed and then the 30-second test.
Quality of life questionnaire | 6 months
  The 36-Item Short Form Survey (SF-36) is an outcome measure instrument that is often used, well-researched, self-reported measure of health. The SF-36 measures eight scales: physical functioning (PF), role physical (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role emotional (RE), and mental health (MH). The results/scores for the entire scale and for each item separately are between 0 and 100.
Quality of life questionnaire | 6 months
  EuroQol-5D (EQ-5D). The EQ-5D descriptive system is a preference-based HRQL measure with one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The 5 dimensions are classified in a score from 1 to 3 and a last question where you rate your health from 0 to 100.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Zaragoza, Zaragoza, Zaragoza, Spain